CLINICAL TRIAL: NCT00006097
Title: CC-1088 Therapy for Chronic Lymphocytic Leukemia: A Phase I/II Trial
Brief Title: Chemotherapy in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Timothy Ernst, MD, Boston Medical Center
Purpose: Treatment
Other Study IDs: CDR0000068104; BUMC-5092; NCI-V00-1603
Record Dates: First submitted 2000-08-03; First posted 2004-05-04 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2001-05

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CC-1088

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of CC-1088 in treating patients who have chronic lymphocytic leukemia that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of CC-1088 in patients with refractory, progressive, B-cell chronic lymphocytic leukemia. II. Determine the response rate to this treatment in these patients.

OUTLINE: Patients receive oral CC-1088 three times a day for 28 days. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 11-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed refractory, progressive, B-cell chronic lymphocytic leukemia Failed prior first line therapy of chlorambucil or fludarabine (or their equivalent) Progressive disease as defined by at least one of the following: Greater than 50% increase in the sum of the products of at least 2 lymph nodes on two consecutive determinations 2 weeks apart (at least one lymph node must be greater than 2 cm) Appearance of new palpable lymph nodes At least a 50% increase in size of previously palpable liver or spleen Appearance of palpable hepatomegaly or splenomegaly not previously present At least a 50% increase in the absolute lymphocyte count to at least 5,000/mm3 Transformation to an aggressive histology (e.g., Richter's or prolymphocytic leukemia) High risk OR Intermediate risk with active disease, as defined by the following: Greater than 10% weight loss Extreme fatigue Fevers greater than 100.5 Fahrenheit for greater than 2 weeks without infection Night sweats Splenomegaly greater than 6 cm Lymphadenopathy greater than 10 cm Lymphocytosis with a doubling time less than 6 months

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG or Zubrod 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) ALT and AST no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception during and for 2 weeks after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Ernst, MD, Study Chair — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States